CLINICAL TRIAL: NCT01285362
Title: Fish Oil for the Treatment of Nonalcoholic Fatty Liver Disease in Children
Brief Title: Fish Oil and Nonalcoholic Fatty Liver Disease (NAFLD) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAF0695
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Fatty Liver Disease; Hepatic Steatosis; Docosahexaenoic Acid; Eicosapentanoic Acid; Omega-3 Fatty Acids; Elevated Transaminases; Fish oil supplements
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish Oil Supplementation (Group A) (Active Comparator): Group A will receive fish oil capsules, containing n3-Fatty Acids, at a dose of 4g/day. Each 1g capsule will contain 465mg of EPA and 375 mg of docosahexaenoic acid (DHA).
  Interventions: Drug: Fish Oil Supplementation
- Placebo Supplementation (Group B) (Placebo Comparator): Group B will receive corn oil in the capsules at the same dose as Group A. The corn oil capsules will appear identical in size and color to the fish oil capsules.
  Interventions: Drug: Placebo Supplementation

INTERVENTIONS:
Drug: Fish Oil Supplementation — Group A will receive fish oil capsules, containing n3-Fatty Acids, at a dose of 4g/day. Each 1g capsule will contain 465mg of EPA and 375 mg of DHA.
  Other Names: Fish Oil Pills
  Arms: Fish Oil Supplementation (Group A)
Drug: Placebo Supplementation — Group B will receive corn oil in the capsules at the same dose as Group A. The corn oil capsules will appear identical in size and color to the fish oil capsules.
  Other Names: Placebo Pills
  Arms: Placebo Supplementation (Group B)

SUMMARY:
Over the past 30 years, the prevalence of childhood obesity in the United States has tripled from 5% to 15%. Major consequences of obesity include insulin resistance, type- 2 diabetes, cardiovascular disease and nonalcoholic fatty liver disease (NAFLD). The liver pathology encompasses a range from isolated fatty liver to advanced fibrosis, cirrhosis and end-stage liver disease. Weight loss, particularly if gradual, may lead to improvement in liver histology. Unfortunately, few patients in the pediatric population are willing to follow these recommendations and achieve weight loss. Medical treatment directed specifically at the liver disease has only recently been investigated and approved in patients with NAFLD. The beneficial effects of fish oil are attributed to its high concentrations of n - 3 fatty acids: eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), which are major regulators of pathways that participate in decreased production and break down of triglycerides and fatty acids in the liver. The investigators hypothesize that children with obesity related NAFLD will normalize elevated liver enzymes, plasma lipid levels, and attenuate insulin resistance with supplements of n-3 fatty acids. If this hypothesis is proven true, then fish oil could be used to treat NAFLD and to prevent the deterioration of fatty liver into end-stage liver disease.

DETAILED DESCRIPTION:
Scientific Abstract:

Over the past 30 years, the prevalence of childhood obesity in the United States has tripled from 5% to 15%. Overweight is defined as a body mass index (BMI) above the 95%centile for age and gender. The recent estimates of obesity prevalence based on the National Health and Nutrition Examination Study (NHANES) 1999-2000 suggest that 15.3% to 15.5% of 6-19 year old children have a BMI above the 95% centile for age. Major consequences of obesity include insulin resistance, type 2 diabetes mellitus, cardiovascular disease and nonalcoholic fatty liver disease (NAFLD). NAFLD represents a spectrum of conditions characterized by macrovesicular hepatic steatosis. The liver pathology encompasses a range from isolated fatty liver to steatohepatitis, advanced fibrosis, cirrhosis and end-stage liver disease. Nonalcoholic steatohepatitis (NASH) may progress to cirrhosis even in children. Weight loss, particularly if gradual, may lead to improvement in liver histology. Unfortunately, few patients in the pediatric population are willing to follow these recommendations and achieve weight loss. Pharmacological therapy directed specifically at the liver disease has only recently been investigated in patients with NAFLD. Most of these studies have been uncontrolled pilot studies, lasting one year or less and have produced equivocal results. Thus, there is currently no effective treatment for this disorder. The beneficial effects of fish oil are attributed to its high concentrations of n - 3 fatty acids: eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). Long-chain polyunsaturated n-3 FA (LCPUFA) are major regulators of molecular pathways altering many areas of cellular and organ function, metabolism and gene expression, and are active in reducing inflammation through the eicosanoid pathway. N-3 LCPUFA are well established negative regulators of hepatic lipogenesis. Recently it has been shown that the suppressive effects of n-3 LCPUFA on lipogenic enzymes are mediated by the reduction of mature SREBP-1c protein in the liver, a key transcription factor that activates transcription of genes involved in fatty acid synthesis. It is also well established today that the n-3 LCPUFA act as PPAR-alpha and gamma modulators, important in triglyceride (TG) and fatty acid catabolism. N-3 LCPUFA produce a dramatic increase in the size and number of hepatic peroxisomes and increase the capacity of the hepatocyte to metabolize fatty acids by inducing peroxisomal beta-oxidation enzymes, such as acyl CoA oxidase . We hypothesize that children with obesity related NAFLD will normalize elevated liver enzymes, plasma lipid levels, and attenuate insulin resistance with supplements of n-3 LCPUFA. If this hypothesis is proven true, then fish oil could be used to treat NAFLD and to prevent the deterioration of fatty liver into end-stage liver disease.

The investigators will study 20 patients with NAFLD and hypertriglyceridemia, age 12y and above. Excluded from the study will be those with evidence of chronic infectious hepatitis, metabolic liver disease, autoimmune and chronic cholestatic liver diseases, insulin dependent diabetes and those with history of alcohol consumption, or exposure to drugs or hepatotoxins. Those qualifying for this study will be age 12 and above obese individuals (BMI > 95% for age), who have hyperlipidemia, but will have normal fasting glucose levels. For inclusion all will have elevation of serum aminotransferases to at least 1.5 times the upper limit of normal for a minimum of 3 months and evidence of fatty liver by abdominal ultrasound and liver biopsy. Patients will be randomized to placebo dummy capsules (controls) or n-3 LCPUFA supplements (Lovaza - GlaxoSmithKline (GSK) Pharmaceuticals, provided free of charge) at a dose of 4gr/day. They will be followed up at 3 and 6 months; monitoring height, weight, BMI, liver enzyme levels (ALT, AST, ALP), bilirubin total and direct, Gamma-glutamyl transferase (GGT), plasma phospholipids, plasma lipids, insulin levels and estimation of HOMA-R.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI i.e. wt(Kg)/ht(m)2) above the 95th % as defined by the NHANES tables.
* Elevated liver enzymes (ALT and/or AST) to at least 1.5 times the upper limit on at least 2 examinations, (ALT, the upper limit of normal values in our laboratory is 41 U/L; AST, upper limit of normal values in our laboratory is 38 U/L).
* Subjects must demonstrate ability to swallow capsules.

Exclusion Criteria:

* Overt Diabetes
* Viral or autoimmune hepatitis, Wilson's disease, Alpha-1 antitrypsin deficiency, hemochromatosis or any other form of chronic liver disease not related to NAFLD
* Exposure to drugs or hepatotoxins less than 14 days prior to recruitment
* Alcohol consumption > 20 grams/day
* Evidence of cirrhosis on liver biopsy.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Martinez, MD, Principal Investigator — Columbia University
Locations (1):
- Irving Clinical Research Center (GCRC) at Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fish Oil Supplementation (Group A): Group A will receive fish oil capsules, containing n3-Fatty Acids, at a dose of 4g/day. Each 1g capsule will contain 465mg of EPA and 375 mg of DHA.
  Fish Oil Supplementation: Group A will receive fish oil capsules, containing n3-Fatty Acids, at a dose of 4g/day. Each 1g capsule will contain 465mg of EPA and 375 mg of DHA.
Period: Overall Study
Arm/Group | Fish Oil Supplementation (Group A) | Placebo Supplementation (Group B)
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil Supplementation (Group A) | Placebo Supplementation (Group B) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16 [14.5 to 16.75] | 15 [13.5 to 15.75] | 15.5 [14.25 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Participants With Normalized Liver Enzyme Levels
Description: To evaluate the number of participants (young adults with obesity related NAFLD) that will normalize their elevated liver enzyme levels (normalized defined as having liver enzyme levels within a normal laboratory range) with supplements of fish oil (n-3 FA containing eicosapentanoic acid and docosahexaenoic acid).
Time Frame: Up to 12 months from entry into the study
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Supplementation (Group A) | Placebo Supplementation (Group B)
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With Normalization of Plasma Lipid Levels
Description: The number of participants (young adults with obesity-related NAFLD and associated dyslipidemia) that will normalize plasma lipid levels (normalized defined as having plasma lipid levels within a normal laboratory range) after fish oil supplementation.
Time Frame: Up to 12 months from entry into the study
Population: Plasma lipid levels were obtained for 6 participants (3 in each group).
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Supplementation (Group A) | Placebo Supplementation (Group B)
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Insulin Resistance Attenuated
Description: The number of participants (young adults with obesity related NAFLD and insulin resistance) that will attenuate insulin resistance (attenuation of insulin resistance defined as decrease in the body's need for insulin and measured by insulin levels and estimation of Homeostatic model assessment (HOMA-R) after fish oil supplementation.
Time Frame: Up to 12 months from entry into the study
Population: Zero participants from group A were analyzed, as insulin levels were not collected at follow-up. Insulin levels were not collected at follow-up as insulin levels were within normal limits at baseline. Two participants in group B were analyzed; 2 of the 4 participants in group B had insulin levels collected at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil Supplementation (Group A) | Placebo Supplementation (Group B)
Number analyzed (Participants) | 0 | 2
Participants |  | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Family and patients were instructed to call with any new symptom, even if minor, after the therapeutic intervention (Group A (active) or group B (placebo)).
Groups:
- Fish Oil Supplementation (Group A): Group A will receive fish oil capsules, containing n3-Fatty Acids, at a dose of 4g/day. Each 1g capsule will contain 465mg of EPA and 375 mg of DHA.
Arm/Group | Fish Oil Supplementation (Group A) | Placebo Supplementation (Group B)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No